CLINICAL TRIAL: NCT02921789
Title: A Phase 2a, Randomized, Open-Label, Active Control, Multi-Center Study to Assess the Efficacy and Safety of Bleselumab in Preventing the Recurrence of Focal Segmental Glomerulosclerosis in de Novo Kidney Transplant Recipients
Brief Title: Study to Assess the Efficacy and Safety of Bleselumab in Preventing the Recurrence of Focal Segmental Glomerulosclerosis in de Novo Kidney Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7163-CL-3201
Record Dates: First submitted 2016-09-30; First posted 2016-10-03 (Estimated); Results first posted 2022-01-05 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Kidney Transplantation; Primary Focal Segmental Glomerulosclerosis (FSGS)
Keywords: Bleselumab; ASKP1240; Efficacy and Safety
MeSH Terms: interventions — bleselumab; Basiliximab; Mycophenolic Acid; Tacrolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) Regimen (Active Comparator): Participants received SOC regimen (basiliximab induction, MMF, Tacrolimus, Methylprednisone, Prednisolone). Basiliximab 20 milligrams (mg) administered by intravenous injection prior to transplantation or intra- operatively before revascularisation as induction therapy and 20mg on day 3 or 4 or 5 post-transplant. MMF 1 gram (g) administered orally or intravenously twice daily until 12 months post transplant. Tacrolimus 0.1 milligram per kilogram per day (mg/kg/day) (two equally divided doses at 0.05 mg/kg/day every 12 hours with a target trough level of 4 - 11 nanogram per milliliter (ng/mL) administered orally within 48 hours post-transplant until 12 months post transplant. Methylprednisone 500, 250, 125 and 60mg administered orally or intravenously on days 0, 1, 2 and 3 respectively and continue through 12 months post transplant. Prednisolone administered orally by tapered doses of 20-30 mg on days 4-14, 10-20mg on days 15-28, 5-10mg on days 29 through 12 months post transplant.
  Interventions: Drug: Basiliximab; Drug: Mycophenolate Mofetil (MMF); Drug: Tacrolimus Capsules; Drug: Methylprednisone; Drug: Prednisone
- Bleselumab Regimen (Experimental): Participants received bleselumab regimen (basiliximab induction, bleselumab, Tacrolimus, Methylprednisone, Prednisolone). Basiliximab 20mg administered by intravenous injection prior to transplantation or intra - operatively before revascularisation as induction therapy and 20mg on day 3 or 4 or 5 post-transplant. Bleselumab 200mg administered by intravenous infusion on day 0, 7, 14, 28, 42, 56, 70, 90 and once per month until month 12. Tacrolimus 0.1 mg/kg/day (two equally divided doses at 0.05 mg/kg/day every 12 hours with a target trough level of 4 - 11 ng/mL) administered orally within 48 hours post transplant until 12 months post transplant. Methylprednisone 500, 250, 125 and 60mg administered orally or intravenously on days 0, 1, 2 and 3 respectively and continue through 12 months post transplant. Prednisolone administered orally by tapered doses of 20-30 mg on days 4-14, 10-20mg on days 15-28, 5-10mg on days 29 through 12 months post transplant.
  Interventions: Drug: Bleselumab; Drug: Basiliximab; Drug: Tacrolimus Capsules; Drug: Methylprednisone; Drug: Prednisone

INTERVENTIONS:
Drug: Bleselumab — Intravenous infusion
  Other Names: ASKP1240
  Arms: Bleselumab Regimen
Drug: Basiliximab — Bolus injection
  Other Names: Simulect®
Drug: Mycophenolate Mofetil (MMF) — Oral Intravenous
  Other Names: CellCept®; MMF
  Arms: Standard of Care (SOC) Regimen
Drug: Tacrolimus Capsules — Oral Capsule
  Other Names: Prograf®
Drug: Methylprednisone — Oral or Intravenous
Drug: Prednisone — Oral Tablet

SUMMARY:
The purpose of this study was to assess the efficacy of the bleselumab regimen (basiliximab induction, tacrolimus, steroids and bleselumab) compared with the Standard of Care (SOC) regimen (basiliximab induction, tacrolimus, steroids and mycophenolate mofetil [MMF]) in the prevention of recurrent Focal Segmental Glomerulosclerosis (rFSGS) defined as nephrotic range proteinuria with protein-creatinine ratio (≥ 3.0 g/g) through 3 months post-transplant. Death, graft loss or lost to follow-up were imputed as rFSGS.

DETAILED DESCRIPTION:
The study consisted of the following periods: Screening (Days -21 to -1), Transplant (Day 0), Post-Transplant (Day 0/post-skin closure through 12 months post-transplant). All subjects entered into a Screening Period (Days -21 to -1 prior to transplant), and underwent a Transplant (Day 0 [zero]), and then followed for up to 12 months in the Post-Transplant Period (Day 0 through 12 months post-transplant).

ELIGIBILITY:
Inclusion Criteria:

* Subject is a recipient of a de novo kidney from a living or deceased donor and has biopsy-proven, primary FSGS (pFSGS) as a cause of end stage renal disease (ESRD) in the subject's native kidneys (initial diagnosing biopsy report is required). A subject who has biopsy-proven pFSGS as a cause of ESRD, and the subject's most current graft failure(s) is due to the recurrence of FSGS, is eligible.
* Subject is anticipated to receive first oral dose of tacrolimus within 48 hours of transplant procedure.
* Subject must be willing and able to comply with the study requirements including prohibited concomitant medication restrictions.
* Subject agrees not to participate in another interventional study while on treatment.

Exclusion Criteria:

* Subject has Induction therapy, other than study-assigned basiliximab, planned as part of initial immunosuppressive regimen.
* Subject has a diagnosis of secondary FSGS (familial, virus associated, medication, etc.) or a defined genetic cause of FSGS.
* Subject has previously received any organ transplant including a kidney and the most current graft failure(s) is not due to the recurrence of FSGS.
* Subject will receive a kidney as part of a multi-organ transplant.
* Subject will receive a dual kidney transplant from a deceased donor.
* Subject will receive a kidney with an anticipated cold ischemia time (CIT) of > 30 hours.
* Subject will receive a kidney that meets BOTH Extended Criteria Donor (ECD) and Donation after Cardiac Death (DCD) criteria. (A kidney that meets either ECD OR DCD criteria may be eligible for inclusion.)
* Subject will receive a blood group system (A, AB, B, O, ABO) incompatible (including A2 into B or O) donor kidney.
* Recipient or donor is known to be seropositive for human immuno-deficiency virus (HIV).
* Subject has a current calculated panel reactive antibody (cPRA) level > 50%.
* Subject has a current malignancy or a history of malignancy (within the past 5 years), except nonmetastatic basal or squamous cell carcinoma of the skin that has been treated successfully, or a renal cell carcinoma that has been treated successfully more than 2 years prior to transplantation.
* Subject has significant liver disease, defined as having during the past 21 days consistently elevated aspartate aminotransferase (AST) (SGOT) and/or alanine aminotransferase (ALT) (SGPT) levels greater than 1.5 times the upper value of the normal range of the investigational site.
* Subject is known to have a positive test for latent tuberculosis (TB) and has not previously received adequate anti-microbial therapy/or would require TB prophylaxis after transplant.
* Subject has an uncontrolled concomitant infection or any other unstable medical condition that could interfere with the study objectives.
* Subject is concurrently participating in another drug study or has received an investigational drug up to 30 days or 5 half-lives prior to transplant.
* Subject is currently receiving or has received up to 8 weeks prior to transplant an immunologic biologic compound (i.e., tumor necrosis factor (TNF) inhibitors, [e.g., etanercept, adalimumab], intravenous immunoglobulin (IVIG)). A subject who has previously received a kidney organ transplant and is currently on an immunosuppression regimen that includes MMF, or any of its components, must discontinue MMF.
* Subject has previously received bleselumab or participated in a clinical study with bleselumab.
* Subject has a known hypersensitivity to tacrolimus, MMF, basiliximab, corticosteroids, or any of the components.
* Subject has any form of substance abuse, psychiatric disorder, or a condition that could invalidate communication with the Investigator.
* Subject has a clinically significant abnormal electrocardiogram (ECG) at Screening.
* Subject is unlikely to comply with the visits scheduled in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (23):
- United States (20):
  - University of Arizona, Tucson, Arizona
  - Stanford School of Medicine, Palo Alto, California
  - UCSF, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Tulane University Health Service Center, New Orleans, Louisiana
  - Michigan Medicine, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - St. Barnabas, Livingston, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania Health System, PCAM, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Utah Medical Center, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
- Canada (3):
  - Site CA15002, Edmonton, Alberta
  - Site CA15005, Vancouver, British Columbia
  - Site CA15006, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Shoji J, Goggins WC, Wellen JR, Cunningham PN, Johnston O, Chang SS, Solez K, Santos V, Larson TJ, Takeuchi M, Wang X. Efficacy and Safety of Bleselumab in Preventing the Recurrence of Primary Focal Segmental Glomerulosclerosis in Kidney Transplant Recipients: A Phase 2a, Randomized, Multicenter Study. Transplantation. 2024 Aug 1;108(8):1782-1792. doi: 10.1097/TP.0000000000004985. Epub 2024 Jul 20. PMID 39042770
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/?pid=7163-CL-3201
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14809&tenant=MT_AST_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across multiple sites in Canada and USA. A total of 67 participants were randomized but 63 participants underwent a kidney transplant and received study drug.
Pre-assignment Details: Male or female participants with ≥ 18 years of age who were recipient of a de novo kidney from a living or deceased donor and has biopsy proven, primary focal segmental glomerulosclerosis (pFSGS) as a cause of ESRD in their native kidneys and their most current graft failure(s) was due to biopsy-proven, recurrent focal segmental glomerulosclerosis (rFSGS).
Period: Overall Study
Arm/Group | Standard of Care (SOC) Regimen | Bleselumab Regimen
Started | 34 | 29
Randomized and Took Study Drug | 34 | 29
Completed | 26 | 25
Not Completed | 8 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Deviation | 2 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Miscellaneous | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety (SAF) population: All participants who were randomized and received at least 1 dose of study drug.
Groups:
- SOC Regimen: Participants received SOC regimen (basiliximab induction, MMF, Tacrolimus, Methylprednisone, Prednisolone). Basiliximab 20mg administered by intravenous injection prior to transplantation or intra- operatively before revascularisation as induction therapy and 20mg on day 3 or 4 or 5 post-transplant. MMF 1g administered orally or intravenously twice daily until 12 months post transplant. Tacrolimus 0.1 mg/kg/day (two equally divided doses at 0.05 mg/kg/day every 12 hours with a target trough level of 4 - 11 ng/mL) administered orally within 48 hours post transplant until 12 months post transplant. Methylprednisone 500, 250, 125 and 60mg administered orally or intravenously on days 0, 1, 2 and 3 respectively and continue through 12 months post transplant. Prednisolone administered orally by tapered doses of 20-30 mg on days 4-14, 10-20mg on days 15-28, 5-10mg on days 29 through 12 months post transplant.
- Bleselumab Regimen: Participants received bleselumab regimen (basiliximab induction, bleselumab, Tacrolimus, Methylprednisone, Prednisolone). Basiliximab 20mg administered by intravenous injection prior to transplantation or intra - operatively before revascularisation as induction therapy and 20mg on day 3 or 4 or 5 post transplant. Bleselumab 200mg administered by intravenous infusion on day 0, 7, 14, 28, 42, 56, 70, 90 and once per month until month 12. Tacrolimus 0.1 mg/kg/day (two equally divided doses at 0.05 mg/kg/day every 12 hours with a target trough level of 4 - 11 ng/mL) administered orally within 48 hours post-transplant until 12 months post transplant. Methylprednisone 500, 250, 125 and 60mg administered orally or intravenously on days 0, 1, 2 and 3 respectively and continue through 12 months post transplant. Prednisolone administered orally by tapered doses of 20-30 mg on days 4-14, 10-20mg on days 15-28, 5-10mg on days 29 through 12 months post transplant.
- Total: Total of all reporting groups
Arm/Group | SOC Regimen | Bleselumab Regimen | Total
Number analyzed (Participants) | 34 | 29 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.9 (13.1) | 41.9 (15.2) | 40.5 (13.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 21 | 18 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 0 | 6
Number of Kidney Transplants [Number; unit: Participants]
  Number of kidney transplants = 1 | 32 | 27 | 59
  Number of kidney transplants = 2 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Recurrence of Focal Segmental Glomerulosclerosis (rFSGS) or Death or Graft Loss or Lost to Follow-up Through 3 Months Post Transplant
Description: rFSGS was defined as nephrotic range proteinuria with a protein/creatinine ratio (≥ 3.0 g/g). Death, graft loss or lost to follow-up was imputed as rFSGS.
Time Frame: At 3 Months post transplant
Population: The Full Analysis Set (FAS) consisted of all participants who are randomized, receive at least one dose of study drug and receive a transplanted kidney. Participants who were later confirmed to have secondary FSGS were excluded from the FAS population because they were not at risk for recurrence post-transplant. Participants with available data at specified time point were included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOC Regimen | Bleselumab Regimen
Number analyzed (Participants) | 32 | 27
Percentage of participants | 31.3 [16.1 to 50.0] | 18.5 [6.3 to 38.1]
Statistical Analysis 1: Comparison: SOC Regimen vs Bleselumab Regimen; Test type: Superiority; p = 0.3705, Fisher Exact — Incidence rate comparisons are based on Fisher's Exact test and confidence intervals are based on Normal Approximation; Difference = -12.7, 95% CI 2-sided [-34.5 to 9.0]

2. Secondary Outcome: Percentage of Participants With rFSGS or Death or Graft Loss or Lost to Follow-up Through 6 and 12 Months Post Transplant
Description: as for outcome 1
Time Frame: At 6 and 12 Months post transplant
Population: FAS population with available data at specified time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOC Regimen | Bleselumab Regimen
Number analyzed (Participants) | 32 | 27
Percentage of participants
  Month 6 | 31.3 [16.1 to 50.0] | 18.5 [6.3 to 38.1]
  Month 12: number analyzed (Participants) | 31 | 26
  Month 12 | 35.5 [19.2 to 54.6] | 23.1 [9.0 to 43.6]
Statistical Analysis 1: Comparison: SOC Regimen vs Bleselumab Regimen; Month 6; Test type: Superiority; p = 0.3705, Fisher Exact — Incidence rate comparisons are based on Fisher's Exact test and confidence intervals are based on Normal Approximation; Difference = -12.7, 95% CI 2-sided [-34.5 to 9.0]
Statistical Analysis 2: Comparison: SOC Regimen vs Bleselumab Regimen; Month 12; Test type: Superiority; p = 0.3890, Fisher Exact — Incidence rate comparisons are based on Fisher's Exact test and confidence intervals are based on Normal Approximation; Difference = -12.4, 95% CI 2-sided [-35.8 to 11.0]

3. Secondary Outcome: Percentage of Participants With Biopsy-Proven Acute Rejection (BPAR) Through 3, 6, and 12 Months Post Transplant
Description: All episodes of kidney dysfunction based on clinical signs and symptoms were evaluated for possible BPAR. BPAR was confirmed if participants Banff criteria >=1.
Time Frame: At 3, 6 and 12 Months post transplant
Population: FAS population with available data at specified time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOC Regimen | Bleselumab Regimen
Number analyzed (Participants) | 30 | 26
Percentage of participants
  Month 3 | 20.0 [7.7 to 38.6] | 26.9 [11.6 to 47.8]
  Month 6 | 20.0 [7.7 to 38.6] | 26.9 [11.6 to 47.8]
  Month 12: number analyzed (Participants) | 29 | 24
  Month 12 | 24.1 [10.3 to 43.5] | 29.2 [12.6 to 51.1]
Statistical Analysis 1: Comparison: SOC Regimen vs Bleselumab Regimen; Month 3; Test type: Superiority; p = 0.7520, Fisher Exact — Incidence rate comparisons are based on Fisher's Exact test and confidence intervals are based on Normal Approximation; Difference = 6.9, 95% CI 2-sided [-15.3 to 29.2]
Statistical Analysis 2: Comparison: SOC Regimen vs Bleselumab Regimen; Month 6; Test type: Superiority; p = 0.7520, Fisher Exact — Incidence rate comparisons are based on Fisher's Exact test and confidence intervals are based on Normal Approximation; Difference = 6.9, 95% CI [-15.3 to 29.2]
Statistical Analysis 3: Comparison: SOC Regimen vs Bleselumab Regimen; Month 12; Test type: Superiority; p = 0.7597, Fisher Exact — Incidence rate comparisons are based on Fisher's Exact test and confidence intervals are based on Normal Approximation; Difference = 5.0, 95% CI 2-sided [-18.9 to 29.0]

4. Secondary Outcome: Percentage of Participants With Efficacy Failure Through 12 Months Post Transplant
Description: Efficacy failure was defined as BPAR, death, graft loss or lost to follow-up through 12 months post transplant.
Time Frame: 12 Months post transplant
Population: FAS Population with available data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOC Regimen | Bleselumab Regimen
Number analyzed (Participants) | 32 | 27
Percentage of participants | 32.3 [16.7 to 51.4] | 32.0 [14.9 to 53.5]
Statistical Analysis 1: Comparison: SOC Regimen vs Bleselumab Regimen; Test type: Superiority; p = 1.0, Fisher Exact — Incidence rate comparisons are based on Fisher's Exact test and confidence intervals are based on Normal Approximation; Difference = -0.3, 95% CI [-24.9 to 24.3]

5. Secondary Outcome: Percentage of Participants With Biopsy Proven rFSGS Through 3, 6 and 12 Months Post-Transplant
Description: Percentage of participants with biopsy-proven rFSGS determined by a blinded central review of images from electron microscopy (EM) and slides for light microscopy (LM) by an independent pathologist.
Time Frame: At 3, 6 and 12 Months post transplant
Population: FAS population with available data at specified time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOC Regimen | Bleselumab Regimen
Number analyzed (Participants) | 30 | 24
Percentage of participants
  Month 3: number analyzed (Participants) | 28 | 22
  Month 3 | 35.7 [18.6 to 55.9] | 31.8 [13.9 to 54.9]
  Month 6: number analyzed (Participants) | 30 | 23
  Month 6 | 36.7 [19.9 to 56.1] | 30.4 [13.2 to 52.9]
  Month 12 | 36.7 [19.9 to 56.1] | 29.2 [12.6 to 51.1]
Statistical Analysis 1: Comparison: SOC Regimen vs Bleselumab Regimen; Month 3; Test type: Superiority; p = 1.0, Fisher Exact — Incidence rate comparisons are based on Fisher's Exact test and confidence intervals are based on Normal Approximation; Difference = -3.9, 95% CI [-30.2 to 22.4]
Statistical Analysis 2: Comparison: SOC Regimen vs Bleselumab Regimen; Month 6; Test type: Superiority; p = 0.7720, Fisher Exact — Incidence rate comparisons are based on Fisher's Exact test and confidence intervals are based on Normal Approximation; Difference = -6.2, 95% CI [-31.7 to 19.3]
Statistical Analysis 3: Comparison: SOC Regimen vs Bleselumab Regimen; Month 12; Test type: Superiority; p = 0.7720, Fisher Exact — Incidence rate comparisons are based on Fisher's Exact test and confidence intervals are based on Normal Approximation; Difference = -7.5, 95% CI [-32.6 to 17.6]

ADVERSE EVENTS:
Time Frame: Day of transplant through 12 months post transplant
Description: SAF population
Arm/Group | SOC Regimen | Bleselumab Regimen
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/29
Serious Adverse Events (participants affected / at risk) | 16/34 | 16/29
Other Adverse Events (participants affected / at risk) | 29/34 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC Regimen (N=34) | Bleselumab Regimen (N=29)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac mass (Cardiac disorders) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 1 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (3) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 5 (6) | 1 (2)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 1 (2)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Polyomavirus-associated nephropathy (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 2 (3) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Exposure via father (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Renal lymphocele (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urine protein/creatinine ratio increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (5) | 2 (2)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 3 (3) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal vein thrombosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 1 (1)
Subclavian steal syndrome (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC Regimen (N=34) | Bleselumab Regimen (N=29)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 8 (9)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 7 (8) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 3 (3)
Vision blurred (Eye disorders) | 2 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (7) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 11 (15) | 8 (9)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (11) | 6 (8)
Vomiting (Gastrointestinal disorders) | 9 (10) | 4 (5)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (5) | 0 (0)
Oedema peripheral (General disorders) | 4 (5) | 5 (5)
Kidney transplant rejection (Immune system disorders) | 1 (1) | 3 (3)
BK virus infection (Infections and infestations) | 3 (3) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 2 (2) | 3 (4)
Escherichia urinary tract infection (Infections and infestations) | 4 (7) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 1 (1)
Polyomavirus viraemia (Infections and infestations) | 5 (7) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 2 (2) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 2 (2)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Incision site pain (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Procedural pain (Injury, poisoning and procedural complications) | 14 (18) | 10 (11)
Alanine aminotransferase increased (Investigations) | 1 (1) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 5 (5)
Blood creatinine increased (Investigations) | 1 (1) | 4 (5)
Histology abnormal (Investigations) | 2 (2) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 2 (2)
Weight increased (Investigations) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Gout (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (9) | 4 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (8) | 6 (7)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (11) | 6 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 9 (10) | 6 (6)
Metabolic acidosis (Metabolism and nutrition disorders) | 7 (9) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 7 (8) | 4 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 11 (12) | 8 (8)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3)
Bladder spasm (Renal and urinary disorders) | 2 (2) | 2 (2)
Dysuria (Renal and urinary disorders) | 3 (3) | 2 (2)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 4 (4) | 1 (1)
Haematuria (Renal and urinary disorders) | 4 (4) | 4 (4)
Oliguria (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 3 (3)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 4 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 5 (5)
Hypotension (Vascular disorders) | 4 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2018-02-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT02921789/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT02921789/SAP_001.pdf